CLINICAL TRIAL: NCT06349317
Title: Neoadjuvant Intensity-modulated Radiotherapy Combined With Perioperative Camrelizumab and Apatinib in the Treatment of Resectable Hepatocellular Carcinoma Associated With Portal Vein Tumor Thrombus: a Single-arm Prospective Clinical Study
Brief Title: Neoadjuvant IMRT Combined With Camrelizumab and Apatinib for Resectable HCC With PVTT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yongyi Zeng (Other)
Responsible Party: Sponsor-Investigator, Yongyi Zeng, Director, Meng Chao Hepatobiliary Hospital of Fujian Medical University
Organization: Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-005
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant intensity-modulated radiotherapy combined with perioperative camrelizumab and apatinib (Experimental): Neoadjuvant intensity-modulated radiotherapy combined with perioperative camrelizumab and apatinib
  Interventions: Combination Product: Neoadjuvant intensity-modulated radiotherapy combined with perioperative camrelizumab and apatinib

INTERVENTIONS:
Combination Product: Neoadjuvant intensity-modulated radiotherapy combined with perioperative camrelizumab and apatinib — 1. Preoperative IMRT targeting PVTT and intrahepatic tumor lesions with a prescribed dose for 18Gy in 6 fractions delivered by using 6-MV X-rays with a linear accelerator at 5 fractions per week;
  2. Perioperative combination of camrelizumab and apatinib Preoperatively, camrelizumab (200mg, every 2 weeks) combined with apatinib (250mg, daily) for 2 cycles (2 weeks as one cycle); Postoperatively, camrelizumab (200mg, every 3 weeks) combined with apatinib (250mg, daily) for 8 cycles (3 weeks as one cycle).

SUMMARY:
This study is an open-label, single-arm prospective clinical trial that evaluates the efficacy and safety of neoadjuvant intensity-modulated radiotherapy combined with perioperative camrelizumab and apatinib in the treatment of resectable hepatocellular carcinoma with portal vein tumor thrombus.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent and able to comply with scheduled visits and related procedures;
2. Age ≥18 and ≤75 years, regardless of gender;
3. Patients with HCC who meet the clinical diagnostic criteria of China's "Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma" (2022 Edition) or are diagnosed by biopsy, and have at least one measurable lesion according to the mRECIST criteria;
4. Presence of portal vein tumor thrombus (PVTT) of Cheng's type I/II/III, with the primary tumor being resectable;
5. Child-Pugh score of Class A;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1;
7. No prior antitumor treatment (such as surgery, radiotherapy, TACE, ablation, chemotherapy, targeted therapy, immunotherapy, or systemic therapy).
8. For patients with hepatitis B virus (HBV) infection, testing for HBV-DNA is required; direct treatment initiation is allowed if HBV-DNA ≤2000 IU/mL; if HBV-DNA >2000 IU/mL, antiviral therapy should be administered for one week before starting the treatment; all HBV positive patients will receive continuous antiviral treatment throughout the study; patients with hepatitis C virus (HCV) RNA positive must undergo antiviral treatment as per the guidelines;
9. Participants must provide a fresh tumor biopsy sample during the screening period (can be waived after discussion with the medical monitor) and blood samples for monitoring immune cells, cytokine levels, and other relevant immune status in the tumor microenvironment;
10. Expected survival of ≥12 weeks;
11. Adequate organ and marrow function, as defined by the following laboratory values:

    1. Hematology: Absolute Neutrophil Count ≥1.5×109/L; Platelets ≥80×109/L; Hemoglobin ≥90g/L;
    2. Liver function: Total bilirubin ≤3× upper limit of normal (ULN); Alanine Aminotransferase and Aspartate Aminotransferase ≤5×ULN; Serum albumin ≥30g/L;
    3. Renal function: Serum creatinine (Cr) ≤1.5×ULN, or for patients with Cr >1.5×ULN, creatinine clearance (CCr) ≥45 mL/min (Cockcroft-Gault formula); Urinalysis showing proteinuria <2+; For participants with baseline proteinuria ≥2+, a 24-hour urine collection and quantitative protein <1g is required;
    4. Coagulation: International Normalized Ratio or APTT ≤1.5×ULN;
12. Females of childbearing potential must agree to abstain from heterosexual intercourse or use effective contraception from signing the informed consent until at least 120 days after the last dose of study medication. They must have a negative serum HCG test within 1 week before treatment and must not be breastfeeding. Females who have not reached menopause (≥12 months of amenorrhea without an alternative medical cause) and have not undergone sterilization (e.g., hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) are considered to be of childbearing potential;
13. Male participants with partners of childbearing potential must agree to abstain from heterosexual intercourse or use reliable and effective contraceptive methods from the time of signing the informed consent until at least 120 days after the last dose of study medication. During the same period, male participants must also agree not to donate sperm. Male subjects whose partners are pregnant must use condoms and do not need to use other contraceptive methods.

Exclusion Criteria:

1. PVTT located in the portal vein branch opposite the tumor, or with inferior vena cava tumor thrombus, extrahepatic metastasis, or tumor invasion of adjacent organs;
2. Known intrahepatic cholangiocarcinoma, sarcomatoid HCC, mixed-cell carcinoma, and fibrolamellar carcinoma; active malignant tumors other than HCC within the past 5 years or concurrently, except for cured localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, and breast carcinoma in situ, which are allowed;
3. Currently with interstitial pneumonia or interstitial lung disease, or history of interstitial lung disease requiring hormone treatment, or other conditions that may interfere with the judgement and management of immunotherapy-related pulmonary toxicity, such as pulmonary fibrosis, organizing pneumonia (e.g., obliterative bronchiolitis), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or participants with active pneumonia or severe impairment of lung function shown on a chest CT during screening; active tuberculosis;
4. Active autoimmune disease or history of autoimmune disease that may recur, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (patients controllable with hormone replacement therapy are allowed); Patients with skin conditions that do not require systemic treatment, such as vitiligo, psoriasis, and alopecia, those with controlled Type I diabetes mellitus undergoing insulin therapy, or individuals whose childhood asthma has fully resolved with no need for intervention in adulthood, are allowed; patients requiring bronchodilators for medical intervention of asthma are not allowed;
5. Use of immunosuppressive drugs or systemic corticosteroids for the purpose of immunosuppression (dose >10mg/day of prednisone or equivalent) within 2 weeks before the start of the study;
6. Active infection, fever of unknown origin ≥38.5°C within 1 week before the study start, or baseline white blood cell count >15×10^9/L; therapeutic antibiotics orally or intravenously within 2 weeks before the study start (excluding prophylactic antibiotics given IV for no more than 48 hours);
7. Congenital or acquired immunodeficiency (e.g., HIV infection);
8. Receipt of live attenuated vaccines within 4 weeks before the study start or expectation of needing such vaccines during the camrelizumab treatment period or within 60 days after the last dose of camrelizuma;
9. Significant bleeding symptoms of clinical significance or a clear bleeding tendency within 6 months before the study start, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, or vasculitis; if baseline fecal occult blood is positive, retesting is allowed, and if still positive, gastroduodenoscopy is required;
10. Known genetic or acquired bleeding (e.g., coagulopathy) and thrombotic tendencies, such as hemophilia, coagulation mechanism disorders, thrombocytopenia, etc.; currently receiving full-dose oral or injectable anticoagulants or thrombolytic agents for therapeutic purposes (prophylactic use of low-dose aspirin, etc., is allowed);
11. Arterial thromboembolic events within 6 months before the study start, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), CTCAE grade 3 or above deep vein thrombosis, pulmonary embolism, etc;
12. Uncontrolled clinical symptoms or diseases of the heart, such as: (1) heart failure of NYHA class II or above or echocardiography showing LVEF <50%; (2) unstable angina; (3) myocardial infarction within 1 year before treatment; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (5) QTc > 450ms for males and >470ms for females (QTc interval calculated using the Fridericia formula; if QTc is abnormal, continuous testing three times at 2-minute intervals is allowed, taking the average value);
13. Hypertension not well controlled with antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg based on the average of ≥2 blood pressure readings), allowing achievement of the above parameters through antihypertensive treatment; history of hypertensive crisis or hypertensive encephalopathy;
14. Major vascular diseases within 6 months before the study start (e.g., requiring surgical repair or recent peripheral arterial thrombosis of an aneurysm);
15. Severe, unhealed, or open wounds and active ulcers or untreated fractures;
16. Major surgery (excluding diagnostic) within 4 weeks before the study start;
17. Inability to swallow pills, malabsorption syndrome, or any condition affecting gastrointestinal absorption;
18. Intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction, including partial obstructions requiring parenteral hydration, parenteral nutrition, or tube feeding related to the underlying disease, within 6 months before the study start. Patients with incomplete obstruction/obstruction syndrome/intestinal obstruction signs/symptoms at initial diagnosis who have undergone definitive (surgical) treatment to alleviate symptoms may be eligible for the study;
19. Use of strong CYP3A4/CYP2C19 inducers, including rifampin (and its analogs) and Hypericum perforatum, or strong CYP3A4/CYP2C19 inhibitors within 2 weeks before the study start;
20. Known allergy to any monoclonal antibody, antiangiogenic targeted drugs, or excipients;
21. Participation in other drug clinical studies within 12 weeks before the study start.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
1-year Event-Free Survival (EFS) rate | 1 year
  EFS is defined as the time from the start of study treatment to the occurrence of tumor progression, relapse assessed by the modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria, death for any reason, or last follow-up (whichever occurs first).

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | up to 2 years
  EFS is defined as the time from the start of study treatment to the occurrence of tumor progression, relapse assessed by the modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria, death for any reason, or last follow-up (whichever occurs first).
Overall Survival (OS) | up to 2 years
  OS is defined as the time from the start of study treatment to death for any reason or the last follow-up (whichever occurs first).
Disease-Free Survival (DFS) | up to 2 years
  DFS is defined as the time from hepatectomy to tumor progression, relapse assessed by mRECIST standards, death for any reason, or last follow-up (whichever occurs first).
R0 resection rate | up to 3 months
  Major Pathological Response, defined as ≤10% viable tumor tissue in the surgical specimen at the time of tumor resection
Overall Objective Response of primary liver tumor and PVTT | up to 3 months
  The assessment of primary liver tumors is consistent with mRECIST criteria; for PVTT, any downstaging in the Cheng's PVTT classification or any conspicuous restoration of blood flow in the portal vein were regarded as partial remission (PR) and any upstaging in the PVTT classification as progressive disease (PD). Otherwise, these outcomes are defined as Stable Disease (SD). If either primary liver tumor or PVTT is classified as PD, the overall response is defined as PD; if either the primary liver tumor or PVTT is PR and the other is SD, it is defined as PR.

OTHER OUTCOMES:
Surgical safety | up to 3 months
  30-day mortality rate post-surgery, surgical complications, reoperation rate, postoperative hospital stay, readmission rate.
Safety of radiotherapy, camrelizumab and apatinib treatment | up to 2 years
  the incidence and severity of adverse events (AE) and serious adverse events (SAE) were determined according to NCI-CTCAE v5.0
Exploratory Endpoints | up to 2 years
  the potential association between changes in the tumor microenvironment and biomarkers with the efficacy of neoadjuvant intensity-modulated radiotherapy combined with perioperative camrelizumab and apatinib treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yongyi Zeng, Professor, Principal Investigator — Meng Chao Hepatobiliary Hospital of Fujian Medical University
Locations (1):
- Mengchao Hepatobiliary Hospital, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No